CLINICAL TRIAL: NCT00996554
Title: Randomized Trial to Compare Two Gastrointestinal Anastomosis Techniques - Single Layer Continuous Versus Double Layer Continuous
Brief Title: Randomized Study Comparing Two Established Gastrointestinal Suture Techniques - One-layer-continuous Versus Double-layer-continuous Suture
Acronym: ANATECH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Feasibility reasons; recruitment was too slow.
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Prof Dr. Stefan Post, Prof. Dr. med., Director of Surgical Department, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK II-MA 0263.5
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Colo-colonic Anastomoses; Ileo-colonic Anastomoses
Keywords: Hand-sutured colo-colonic and ileo-colonic anastomoses in elective surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Double-Layer-Suture (Experimental): Hand-sutured end-to-end or end-to-side anastomosis performed by double-layer continuous technique (monofil thread)
  Interventions: Procedure: double layer-suture
- Single-layer suture (Active Comparator): Hand-sutured end-to-end or end-to-side anastomosis performed by single-layer continuous technique (monofil thread).
  Interventions: Procedure: Single-layer suture

INTERVENTIONS:
Procedure: double layer-suture — Hand-sutured end-to-end or end-to-side anastomosis performed by double-layer continuous technique (monofil thread)
  Arms: Double-Layer-Suture
Procedure: Single-layer suture — Hand-sutured end-to-end or end-to-side anastomosis performed by single-layer continuous technique (monofil thread)
  Arms: Single-layer suture

SUMMARY:
The purpose of this study is to examine the frequency of postoperative complications depending on the number of suture layers in colo-colonic and ileo-colonic anastomoses Hypothesis: double-layer suture has less anastomotic leakages compared to single-layer suture.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old,
* planned for elective surgery
* at least one hand-sutured ileo-colonic or colo-colonic anastomosis

Exclusion Criteria:

* ASA-Score > 3,
* missing written consent of the informed patient
* no existing choice between suture-techniques according to the surgeon
* patient not able to cooperate/non-compliance
* rectal anastomoses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2004-01; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Frequency of clinical anastomostic leaks | 3 months

SECONDARY OUTCOMES:
death of any cause within 3 months post-operatively | 3 months
  all causes of death will be recorded independently of a possible causal relationship with the operation
postoperative morbidity | 30 days
Duration of anastomosis (min) | 1-3 hours
Frequency of anastomotic strictures | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Post, Prof, MD, Principal Investigator — University Medical Center Mannheim, Germany, Surgical Department
Locations (1):
- University Medical Center Mannheim, Surgical Department, Mannheim, Germany

REFERENCES:
- [Background] Herrle F, Diener MK, Freudenberg S, Willeke F, Kienle P, Boenninghoff R, Weiss C, Partecke LI, Schuld J, Post S. Single-Layer Continuous Versus Double-Layer Continuous Suture in Colonic Anastomoses-a Randomized Multicentre Trial (ANATECH Trial). J Gastrointest Surg. 2016 Feb;20(2):421-30. doi: 10.1007/s11605-015-3003-0. Epub 2015 Nov 2. PMID 26525206